CLINICAL TRIAL: NCT02433041
Title: Baden PRIDe Trial - Baden Prevention and Reduction of Incidence of Postoperative Delirium Trial
Brief Title: Baden Prevention and Reduction of Incidence of Postoperative Delirium Trial
Acronym: PRIDe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013DR4089
Record Dates: First submitted 2015-04-07; First posted 2015-05-04 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; Cortisol; NSE; S-100beta; MMSE; Nu-DESC; ICDSC; DOS; Haloperidol; Ketamine; Combination of Haloperidol and Ketamine; Placebo; Prevention of
MeSH Terms: conditions — Emergence Delirium | interventions — Haloperidol; Ketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Haloperidol (Active Comparator): Haloperidol 0.005mg/kg at induction of anesthesia
  Interventions: Drug: Haloperidol
- Ketamine (Active Comparator): Ketamine 1mg/kg at induction of anesthesia
  Interventions: Drug: Ketamine
- Haloperidol + Ketamine (Active Comparator): Combination of Haloperidol + Ketamine in same dosage at induction of anesthesia
  Interventions: Drug: Haloperidol + Ketamine
- Saline solution (NaCl 0.9%) (Placebo Comparator): Placebo
  Interventions: Drug: Saline solution (NaCl 0.9%)

INTERVENTIONS:
Drug: Haloperidol — Haloperidol 0.005mg/kg at induction of anesthesia
  Arms: Haloperidol
Drug: Ketamine — Ketamine 1mg/kg at induction of anesthesia to test its power to prevent postoperative delirium
  Arms: Ketamine
Drug: Haloperidol + Ketamine — Haloperidol 0.005mg/kg + Ketamine 1mg/kg at induction of anesthesia to test their power to prevent postoperative delirium if given together
  Arms: Haloperidol + Ketamine
Drug: Saline solution (NaCl 0.9%) — Placebo being used in one of the four groups
  Arms: Saline solution (NaCl 0.9%)

SUMMARY:
The purpose of this study is to find out whether postoperative delirium can be more properly prevented by the combination of determined preventive agents in past studies. Further on the investigators measure pre- and postoperative cortisol, neuron specific enolase (NSE) and S-100beta levels.

DETAILED DESCRIPTION:
The postoperative delirium remains a challenge for medical stuff concerning detection, therapy and avoidance of consequences. Over the years numerous risk factors were detected which emphasizes the importance of its prevention. Within these studies some possibilities, but no strictly defined rules of action for pharmacological or neuropsychological prevention are described. This is why in this randomized, double-blinded, placebo-controlled study, the investigators want to compare two agents that were found to prevent postoperative delirium to a certain level, even in combination: the investigators arrange the patients within four study groups, one receiving Haloperidol, one Ketamine, one both and one placebo. The patients receive the study drug only once right before induction of anesthesia. After the day of recruitment there is the day of operation and a follow-up of three days (5 days of observation in total, where the investigators will test cognitive function with Mini Mental Status Examination (MMSE), Delirium Observation Scale (DOS), Nursing Delirium Screening Scale (Nu-DESC) or Intensive Care Delirium Screening Checklist (ICDSC). Additionally the investigators will measure and compare pre- and postoperative Cortisol, NSE and S-100beta levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Signed agreement

Exclusion Criteria:

* Delirium at admittance or MMSE score <24 points
* High risk for postoperative ICU treatment
* Haloperidol or Ketamine intolerance
* Risk of lack of cooperation
* Drug an alcohol abuse
* Dementia
* QT interval (QTc) prolongation (at least 460ms in men, at least 470ms women) or drugs influencing QT interval, such as class Ia and III antiarrhythmics, Gatifloxacin, Moxifloxacin, Pentamidin, Cotrimoxazol, Tacrolimus, Dolasetron
* Parkinson's disease
* Intake of dopaminergic drugs (Levodopa, dopamine agonists)
* Parkinsonism
* Epilepsy
* Unable to be interviewed (severe Dementia, speaking disorders, intubation, respiratory isolation, aphasia, coma, terminal illness)
* Delay of operation of more than 72 hours past hospital admittance
* Body weight >100kg

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Differences among study groups - Significant drop in MMSE of two points in one of the three postoperative follow-up days | 5 day follow-up (preoperative, day of surgery, postoperative days 1-3)
  Significant drop in MMSE of two points in one of the three postoperative follow-up days (ICU patients excluded)

SECONDARY OUTCOMES:
Quantification of incidence of postoperative delirium based on cognitive testing and lab parameters | 5 day follow-up (preoperative, day of surgery, postoperative days 1-3)
  Drop of one point in Nursing Delirium Screening Scale (Nu-DESC) compared pre- and postoperatively, comparison of levels of NSE, S-100beta and Cortisol (significantly elevated postoperatively?)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Hollinger, MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Hollinger A, Rust CA, Riegger H, Gysi B, Tran F, Brugger J, Huber J, Toft K, Surbeck M, Schmid HR, Rentsch K, Steiner L, Siegemund M. Ketamine vs. haloperidol for prevention of cognitive dysfunction and postoperative delirium: A phase IV multicentre randomised placebo-controlled double-blind clinical trial. J Clin Anesth. 2021 Feb;68:110099. doi: 10.1016/j.jclinane.2020.110099. Epub 2020 Oct 22. PMID 33120302
- [Derived] Riegger H, Hollinger A, Seifert B, Toft K, Blum A, Zehnder T, Siegemund M. Baden Prevention and Reduction of Incidence of Postoperative Delirium Trial (PRIDe): a phase IV multicenter, randomized, placebo-controlled, double-blind clinical trial of ketamine versus haloperidol for prevention of postoperative delirium. Trials. 2018 Feb 26;19(1):142. doi: 10.1186/s13063-018-2498-6. PMID 29482596